CLINICAL TRIAL: NCT02235987
Title: A Study of the Effect of Ascending Single Doses of DG3173 and 300 μg of Octreotide on Human Growth Hormone Levels in Untreated Acromegalics.
Brief Title: Single Dose Pharmacology Study of DG3173 and Octreotide in Acromegalic Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aspireo Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DG3173-II-01
Record Dates: First submitted 2014-08-14; First posted 2014-09-10 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-01

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — Octreotide; PTR 3173

ARMS (1):
- Octreotide, then ascending DG3173 (Other): Interventions: octreotide and DG3173. Eligible patients are to receive 300 µg octreotide as active comparator, followed by four ascending doses of 100 µg, 300 µg, 900 µg and 1800 µg DG3173. All treatments will be administered consecutively to all patients as single subcutaneous bolus injections.
  Interventions: Drug: octreotide; Drug: DG3173

INTERVENTIONS:
Drug: octreotide — Eligible patients are to receive 300 µg octreotide as active comparator, followed by four ascending doses of 100 µg, 300 µg, 900 µg and 1800 µg DG3173. All treatments will be administered consecutively to all patients as single subcutaneous bolus injections.
Drug: DG3173 — Eligible patients are to receive 300 µg octreotide as active comparator, followed by four ascending doses of 100 µg, 300 µg, 900 µg and 1800 µg DG3173. All treatments will be administered consecutively to all patients as single subcutaneous bolus injections.

SUMMARY:
The study is designed to investigate the safety, tolerability and efficacy of DG3173 in untreated acromegaly patients. Twenty patients received ascending single doses of DG3173 and one dose of octreotide, the current gold standard of medical therapy for acromegaly, with each patient receiving all doses of DG3173 as well as octreotide.

ELIGIBILITY:
Inclusion Criteria:

* Men, women of non childbearing potential or women of child bearing potential who either abstain from sexual intercourse, have a sterile partner or practice a medically approved double barrier method of contraception
* Diagnosis of acromegaly of pituitary origin
* Have age adjusted Insulin like Growth Factor 1 (IGF-1) concentrations ≥1.5 times the upper limit of normal range on two consecutive measurements in the 6 months prior to the first dosing day (including the measurement to be made at screening [Visit 2])
* Have a random hGH level of ≥5 µg/L in the 6 months prior to or at screening (Visit 2)
* Have given written informed consent
* Ability to comply with the requirements of the protocol of the study

Exclusion Criteria:

* Previous specific treatment for acromegaly in the 6 months prior to screening (Visit 2), including somatostatin analogues (SSAs), surgery, radiotherapy and pegvisomant
* Treatment with dopamine agonists in the 3 months prior to screening (Visit 2)
* Uncontrolled hypertension or orthostatic hypotension
* Type I diabetes mellitus, poorly-controlled type II diabetes mellitus (glycosylated haemoglobin [HbA1c]≥7.5%) and patients requiring insulin treatment
* Gallstones or gravel that could cause biliary obstruction
* Hyperprolactinaemia
* Participation in a clinical study within 60 days prior to screening (Visit 2)
* Receipt of blood, blood products or plasma derivatives 60 days prior to screening (Visit 2)
* Pregnancy or lactation
* A history of active alcohol abuse or drug addiction
* Positive viral serology screening result for hepatitis B surface antigen, antibodies to hepatitis C virus, or human immunodeficiency virus type 1 and 2
* Evidence or suspicion of tumour expansion
* Clinically significant abnormality in screening ECG
* Any clinically significant abnormal laboratory safety test (biochemistry, haematology and dipstick urinalysis) in the opinion of the Investigator
* Any disease which in the Investigator's opinion would exclude the patient from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2014-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Octreotide, Then Ascending DG3173
Started | 20
Received Octreotide | 20
Received 100 µg DG3173 | 20
Received 300 µg DG3173 | 20
Received 900 µg DG3173 | 19
Received 1800 µg DG3173 | 19
Completed | 19
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Cross-over: Interventions: octreotide and DG3173. Eligible patients are to receive 300 µg octreotide as active comparator, followed by four ascending doses of 100 µg, 300 µg, 900 µg and 1800 µg DG3173. All treatments will be administered consecutively to all patients as single subcutaneous bolus injections.
Arm/Group | Cross-over
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 2
Region of Enrollment [Number; unit: participants]
  Ukraine | 20

OUTCOME MEASURES:

1. Primary Outcome: Participants With Trough Human Growth Hormone < 2.5 ug/mL
Time Frame: Pre dose and 0.33, 0.67 hours and 1, 1.5, 2, 3, 4, 5, 6 and 8 hours post dose on each dosing day.
Population: Baseline: an 8 hour untreated human growth hormone (hGH) profile was obtained in the period between 15 and 7 days prior to the first study treatment administration.
Measure: Number; unit: participants with trough hGH < 2.5 µg/mL
Arm/Group | Baseline (Untreated Control) | 300 µg Octreotide | 100 µg DG3173 | 300 µg DG3173 | 900 µg DG3173 | 1800 µg DG3173
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 19 | 19
participants with trough hGH < 2.5 µg/mL | 1 | 8 | 4 | 6 | 7 | 8

ADVERSE EVENTS:
Arm/Group | 300 µg Octreotide | 100 µg DG3173 | 300 µg DG3173 | 900 µg DG3173 | 1800 µg DG3173
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 1/20 | 0/20 | 1/20 | 0/19 | 1/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 300 µg Octreotide (N=20) | 100 µg DG3173 (N=20) | 300 µg DG3173 (N=20) | 900 µg DG3173 (N=19) | 1800 µg DG3173 (N=19)
abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Hyperamylasemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No